CLINICAL TRIAL: NCT02301364
Title: A Phase II Trial Of Buparlisib (BKM120) In Patients With Recurrent/Refractory Primary Central Nervous System Lymphoma (PCNSL) and Recurrent/Refractory Secondary Central Nervous System Lymphoma (SCNSL)
Brief Title: Buparlisib (BKM120) In Patients With Recurrent/Refractory Primary Central Nervous System Lymphoma (PCNSL) and Recurrent/Refractory Secondary Central Nervous System Lymphoma (SCNSL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-177
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-02

CONDITIONS: Lymphoma; Primary Central Nervous System Lymphoma; Recurrent/Refractory Secondary Central Nervous System Lymphoma
Keywords: Buparlisib (BKM120); 14-177
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — NVP-BKM120

ARMS (1):
- Buparlisib (BKM120) (Experimental): This is an open-label, phase II trial of the pan-PI3K inhibitor buparlisib (BKM120) for patients with recurrent or refractory primary central nervous lymphoma (PCNSL) and recurrent or refractory secondary central nervous lymphoma (SCNSL).
  Interventions: Drug: Buparlisib (BKM120)

INTERVENTIONS:
Drug: Buparlisib (BKM120) — Buparlisib 100 mg once daily.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, Buparlisib (also known as BKM120) has on lymphoma and the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to understand and be willing to sign a written informed consent document.
* Subjects must be at least 18 years of age on the day of consenting to the study.
* Histologically documented PCNSL or SCNSL. Patients with SCNSL need to have cytology or tissue biopsy documenting lymphomatous involvement of the CNS
* Patients must have relapsed/refractory PCNSL or relapsed/refractory SCNSL
* All patients need to have received at least one prior CNS directed therapy. There is no restriction on the number of recurrences.
* Patients with parenchymal lesions must have unequivocal evidence of disease progression on imaging (MRI of the brain or head CT) 21 days prior to study registration. For patients with leptomeningeal disease only, CSF cytology must document lymphoma cells and/or imaging findings consistent with CSF disease 21 days prior to study registration.
* Participants must have a Karnofsky performance status (KPS) of ≥ 50.
* Participants must have adequate bone marrow and organ function shown by:

Absolute neutrophil count (ANC) ≥ 1.5x 109/L

* Platelets ≥ 100 x 109/L and no platelet transfusion within the past 14 days prior to study registration
* Hemoglobin (Hgb) ≥ 9 g/dL and no red blood cell (RBC) transfusion within the past 14 days prior to study registration
* International Normalized Ratio (INR) ≤ 1.5
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 times the ULN.
* Serum bilirubin ≤ upper limit of normal; or total bilirubin ≤ 2.0x the ULN with direct bilirubin within the normal range in patients with well documented Gilbert Syndrome.

  * Participants must be able to take oral medication.
  * Patients must be able to tolerate MRI scans.
  * Patients must be able to tolerate lumbar puncture and/or Ommaya taps.
  * Participants must have recovered to grade 1 toxicity from prior therapy.
  * Participates must be able to submit 20 unstained slides from the initial tissue diagnosis for confirmation of diagnosis and correlative studies
  * Life expectancy of > 3 months (in the opinion of the investigator) Note: Prior autologous stem cell transplant as well as radiation to the CNS is NOT an exclusion criterion. Prior allogenic stem cell transplant IS an exclusion criterion.

Exclusion Criteria:

* Patients with SCNSL actively receiving treatment for extra-CNS disease are excluded. Patient should have complete resolution of their systemic disease not requiring additional systemic therapy (e.g. maintenance rituximab or decadron).
* The patient has received prior treatment with a PI3K inhibitor, AKT inhibitor, or mTOR inhibitor (e.g. rapamycin, MK2206, perifosine, etc.).
* Patient is concurrently using other approved or investigational antineoplastic agents
* Patient has received chemotherapy or targeted anticancer therapy, monoclonal antibodies ≤ 4 weeks or 5 half-lives, whichever is shorter, or 6 weeks for nitrosourea or mitomycin-C prior to starting the study drug, or the patient has not recovered side the side effects of such therapy
* Patient who has received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered to grade 1 or better from related side effects of such therapy (except alopecia)
* Patient requires more than 8 mg of dexamethasone daily or the equivalent
* Patient is taking an enzyme inducing anti-epileptic drug (EIAED), including phenobarbital, phenytoin, fosphenytoin, primidone, carbamazepine, oxcarbazepine, eslicarbazepine, rufinamide, and felbamate. Participates must be off of any EIAED for a least two weeks prior to starting the study drug
* Patient is taking a drug known to be a strong inhibitor or inducers of the isoenzyme CYP3A. Participants must be off a strong CYP3A inhibitors and inducers for at least two weeks prior to starting the study drug.
* Patient is taking a drug with known risk to promote QT prolongation and Torsade de Pointes Patient is currently using herbal preparations or medications. Participants should stop using herbal medications 7 days prior to the first dose of the study drug.
* Patient is using warfarin or any other Coumadin-derivative anticoagulant. Patients must be off Coumadin-derivative anticoagulants for at least seven days prior to starting the study drug. Low molecular weight heparin is allowed
* Patient has a history of allergic reactions to compounds of similar chemical or biological composition to buparlisib
* Patient has an uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, chronic liver disease, chronic renal disease, pancreatitis, chronic pulmonary disease, or psychiatric illness or social situations that would limit compliance with the study requirements
* Patient has acute viral hepatitis or a history of chronic or active HBV or HCV infection
* Patient has an active concurrent malignancy requiring active therapy.
* Patient is known to have human immunodeficiency virus (HIV) infection
* Patient has any severe psychiatric disease that would interfere with participation in the trial as determined by the study investigator
* Patient has ≥ CTCAE grade 3 anxiety
* Patient has ≥ CTCAE grade 2 diarrhea Patient has a score ≥12 on the PHQ-9 questionnaire
* Patient selects a response of "1, 2 or 3" to question number 9 on the PHQ-9-questionaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9).
* Patient has a GAD-7 mood scale score ≥15.
* Patient has a medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others).
* Patient has active cardiac disease or cardiac dysfunction including any of the following:
* Left ventricular ejection fraction (LVEF) ,50% as determined by Multiple Gated Acquisition (MUGA) scan or echocardiogram (ECHO)
* QTc>480msec on screening ECG (using the QTcF formula)
* Angina pectoris that requires the use of anti-anginal medications
* Ventricular arrhythmias except for benign premature ventricular contractions
* Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
* Conduction abnormality requiring a pacemaker
* Valvular disease with documented compromise in cardiac function
* Symptomatic pericarditis
* Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall motion abnormalities on assessment of left ventricular ejection fraction function
* History of documented congestive heart failure (New York Heart Association functional classification III-IV)
* Documented cardiomyopathy
* Congenital long QT syndrome
* Patient is currently receiving treatment with QT prolonging medication known to have a risk to induce Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
* Patient has impaired gastrointestinal function or gastrointestinal disease affecting absorption of buparlisib (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or extensive small bowel resection).
* Patient has poorly controlled diabetes mellitus with a glycosylated hemoglobin >8% or poorly controlled steroid-induced diabetes mellitus with a glycosylated hemoglobin of >8%.
* Patient underwent major systemic surgery ≤ 2 weeks prior to starting the trial treatment or who has not recovered from the side effects of such surgery.
* Women who are pregnant or nursing (lactating), where pregnancy is defined as a state of a female after conception until the termination of gestation, confirmed by a positive serum hCG laboratory test of > 5 mIU/mL.
* Patients who have received allogenic stem cell transplants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-11-20; Primary Completion 2016-10-11 (Actual); Study Completion 2016-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grommes, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Grommes C, Pentsova E, Schaff LR, Nolan CP, Kaley T, Reiner AS, Panageas KS, Mellinghoff IK. Preclinical and clinical evaluation of Buparlisib (BKM120) in recurrent/refractory Central Nervous System Lymphoma. Leuk Lymphoma. 2023 Sep;64(9):1545-1553. doi: 10.1080/10428194.2023.2223734. Epub 2023 Jun 15. PMID 37317993
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 11/20/2014 Protocol Closed to Accrual 03/22/2/016 Primary Completion Date 10/11/2016 Recruitment Location is the medical clinic
Period: Overall Study
Arm/Group | Buparlisib (BKM120)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Buparlisib (BKM120)
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 64 [55 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the time from the date of treatment start to the date of the first documented PD or death due to any cause. PFS will be based on the investigator's assessment of MRI, CSF studies and clinical presentation.
Time Frame: 2 years
Measure: Median (Full Range); unit: days
Arm/Group | Buparlisib (BKM120)
Number analyzed (Participants) | 4
days | 39 [30 to 78]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events be summarized based on the Common Toxicity Criteria version 4.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Buparlisib (BKM120)
Number analyzed (Participants) | 4
Participants | 4

3. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from treatment start to the date of death due to any cause.
Time Frame: 2 years
Measure: Median (Full Range); unit: days
Arm/Group | Buparlisib (BKM120)
Number analyzed (Participants) | 4
days | 196 [54 to 284]

4. Secondary Outcome: Overall Response Rate
Description: This study will use the Macdonald criteria. Specific lesions must be evaluated serially, and comparative analysis of changes in the area of contrast enhancement, as well as the non-enhancing component, should be performed. Complete Response: Complete disappearance of all measurable and non-measurable disease. No new lesions. Partial Response: Great than or equal to 50% decrease over the baseline in the sum of products of perpendicular diameters of all measurable lesions. no progression of non-measurable disease. No new lesions. Stable/No Response: Does not qualify for CT, PR, or progression. Progressive Disease: 25% increase in the sum of products of all measureable lesions over smallest sum observes (or baseline if no decrease), OR clear clinical worsening of any non-measurable disease, OR appearance of any new lesion/site, OR clear clinical worsening or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Buparlisib (BKM120)
Number analyzed (Participants) | 4
Participants
  Partial Response | 1
  Progressive Disease | 3

ADVERSE EVENTS:
Time Frame: Up to 30 days post treatment
Arm/Group | Buparlisib (BKM120)
All-Cause Mortality (participants affected / at risk) | 3/4
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buparlisib (BKM120) (N=4)
Confusion (Psychiatric disorders) | 1
Death NOS (General disorders) | 1
Depression (Psychiatric disorders) | 1
Dysphasia (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Buparlisib (BKM120) (N=4)
Anemia (Blood and lymphatic system disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4
Platelet count decreased (Investigations) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
INR increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Cognitive disturbance (Nervous system disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Lymphocyte count decreased (Investigations) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
White blood cell decreased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Cholesterol high (Investigations) | 1
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysphasia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Fatigue (General disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Seizure (Nervous system disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT02301364/Prot_SAP_000.pdf